CLINICAL TRIAL: NCT00171041
Title: A Double-Blind, Randomized, Multi-Center Study Followed By 12 Months Open-Label Treatment To Evaluate The Dose Response And Safety Of Valsartan In Pediatric Hypertensive Patients
Brief Title: A Study Of Valsartan Used To Treat Hypertension For Up To 13 Months In Hypertensive Children Ages 6 - 16 Years Of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2302
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: PEDIATRIC HYPERTENSION; PEDIATRIC; VALSARTAN
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
Drugs used to treat high blood pressure in adults should also be effective in treating high blood pressure in children and adolescents. This study will test the safety and efficacy of valsartan in treating high blood pressure in hypertensive children 6-16 years of age whose parent(s)/guardian(s) grant permission to participate.

ELIGIBILITY:
Inclusion Criteria:

* CHILDREN HAVE SYSTOLIC BLOOD PRESSURE AT A LEVEL =>95th PERCENTILE FOR AGE/GENDER/HEIGHT
* CONSENT FROM PARENT(S)/GUARDIAN(S) MUST BE GRANTED

Exclusion Criteria:

* BLOOD PESSURE IS =>5% HIGHER THAN 99th PERCENTILE FOR AGE
* SERIOUS, CLINICALLY SIGNIFICANT FINDINGS UPON PHYSICAL EXAMINATION, AND LABORATORY AND OTHER ASSESSMENTS

Other protocol-defined inclusion/exclusion criteria will also apply.

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 265 (Actual)
Dates: Start 2002-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic blood pressure after 2 weeks

SECONDARY OUTCOMES:
Change from baseline systolic and diastolic blood pressure after 4 weeks and 52 weeks
Change from baseline systolic blood pressure after 4 weeks
Change from baseline diastolic blood pressure after 2 weeks
Change in diastolic blood pressure after 2 weeks to 4 weeks
Change from baseline diastolic blood pressure after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, E.Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Wells T, Blumer J, Meyers KE, Neto JP, Meneses R, Litwin M, Vande Walle J, Solar-Yohay S, Shi V, Han G; Valsartan Pediatric Hypertension Study Group. Effectiveness and safety of valsartan in children aged 6 to 16 years with hypertension. J Clin Hypertens (Greenwich). 2011 May;13(5):357-65. doi: 10.1111/j.1751-7176.2011.00432.x. Epub 2011 Mar 18. PMID 21545397